CLINICAL TRIAL: NCT00777946
Title: A Randomized, Eight-week Double-blind, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren / Amlodipine (300/5 mg and 300/10 mg) in Comparison With Aliskiren 300 mg in Patients With Essential Hypertension Not Adequately Responsive to Aliskiren 300 mg Monotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of Combination Aliskiren/Amlodipine in Patients Not Adequately Responding to Aliskiren Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100A2303
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Aliskiren, Amlodipine, Non-responder to aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aliskiren 300 mg/Amlodipine 5 mg (Experimental): Participants received 1 Aliskiren/Amlodipine 300/5mg tablet + 1 Placebo to Aliskiren tablet once daily in the morning for 8 weeks.
  Interventions: Drug: Aliskiren/Amlodipine 300/5 mg; Drug: Placebo to Aliskiren
- Aliskiren 300 mg/Amlodipine 10 mg (Experimental): Participants received 1 Aliskiren/Amlodipine 300/10 mg tablet + 1 Placebo to Aliskiren tablet orally once daily in the morning for 8 weeks.
  Interventions: Drug: Aliskiren/Amlodipine 300/10 mg; Drug: Placebo to Aliskiren
- Aliskiren 300 mg (Active Comparator): Participants received 1 Aliskiren 300 mg tablet + 1 Placebo to Aliskiren/Amlodipine tablet orally once daily in the morning for 8 weeks.
  Interventions: Drug: Aliskiren 300 mg; Drug: Placebo to Aliskiren/Amlodipine

INTERVENTIONS:
Drug: Aliskiren 300 mg — Aliskiren 300 mg tablet taken orally once a day with a glass of water.
  Arms: Aliskiren 300 mg
Drug: Aliskiren/Amlodipine 300/5 mg — Aliskiren/Amlodipine 300/5 mg tablet taken orally once a day with a glass of water.
  Arms: Aliskiren 300 mg/Amlodipine 5 mg
Drug: Aliskiren/Amlodipine 300/10 mg — Aliskiren/Amlodipine 300/10 mg taken orally once a day with a glass of water.
  Arms: Aliskiren 300 mg/Amlodipine 10 mg
Drug: Placebo to Aliskiren — Placebo to Aliskiren tablet taken orally once a day.
  Arms: Aliskiren 300 mg/Amlodipine 10 mg; Aliskiren 300 mg/Amlodipine 5 mg
Drug: Placebo to Aliskiren/Amlodipine — Placebo to Aliskiren/Amlodipine taken orally once a day.
  Arms: Aliskiren 300 mg

SUMMARY:
This study will assess the safety and efficacy of combination aliskiren/amlodipine in patients not adequately controlled with aliskiren alone

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients or patients who have not been treated for hypertension within the 4 weeks prior to Visit 1 must have a mean sitting Diastolic Blood Pressure (msDBP) ≥ 95 mmHg and < 110 mmHg at Visits 1 and 2
* Patients who have been treated for hypertension within the 4 weeks prior to - Visit 1 must have a msDBP ≥ 90 mmHg and < 110 mmHg at Visit 2
* All patients must have a msDBP ≥ 90 mmHg and < 110 mmHg at Visit 4

Exclusion Criteria:

* Severe hypertension
* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* Previous or current diagnosis of heart failure New York Heart Association (NYHA Class II-IV)
* Serum potassium ≥ 5.3 mEq/L (mmol/L) at Visit 1
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Hypersensitivity to renin inhibitors, calcium channel blockers, or to drugs with Similar chemical structures
* History of hypertensive encephalopathy or cerebrovascular accident, or history of transient ischemic attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (9):
- Investigative site, Estonia, Estonia
- Investigative site, France, France
- Investigative Site, Iceland, Iceland
- Investigative Site, India, India
- Investigative site, Italy, Italy
- Investigative Site, Lithuania, Lithuania
- Investigative Site, Republic of Korea, South Korea
- Investigative Site, Spain, Spain
- Investigative Site, Venezuela, Venezuela

REFERENCES:
- [Derived] Glorioso N, Thomas M, Troffa C, Argiolas G, Patel S, Baek I, Zhang J. Antihypertensive efficacy and tolerability of aliskiren/amlodipine single- pill combinations in patients with an inadequate response to aliskiren monotherapy. Curr Vasc Pharmacol. 2012 Nov;10(6):748-55. doi: 10.2174/157016112803520765. PMID 22303910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 7 day wash-out period and a 4 week single-blind run-in period prior to the 8 week double-blind period.
  2 of the 820 randomized patients were randomized in error, are not included in the 818 participants enrolled in the double-blind period, did not receive study drug & are not included in the Safety and Full Analysis Sets.
Groups:
- Aliskiren 300 mg/Amlodipine 10 mg: Participants received 1 Aliskiren/Amlodipine 300/10mg tablet + 1 Placebo to Aliskiren tablet once daily in the morning for 8 weeks.
Period: Overall Study
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Started | 283 (1 patient in the Aliskiren 300 mg/Amlodipine 10 mg group was randomized in error.) | 277 (1 patient in the Aliskiren 300 mg/Amlodipine 5 mg group was randomized in error.) | 260
Safety & Full Analysis Sets | 282 | 276 | 260
Completed | 262 | 271 | 244
Not Completed | 21 | 6 | 16
Not completed — Adverse Event | 11 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 9
Not completed — Condition no longer required study drug | 1 | 0 | 0
Not completed — Patient withdrew consent | 3 | 2 | 3
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Protocol deviation | 2 | 1 | 1
Not completed — Randomized in error | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg | Total
Number analyzed (Participants) | 283 | 277 | 260 | 820
Age Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.67) | 54.4 (10.69) | 54.7 (10.99) | 54.6 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 101 | 103 | 324
  Male | 163 | 176 | 157 | 496

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study in the Mean Sitting Diastolic Blood Pressure (msDBP)
Description: After the patient had been sitting for 5 minutes, systolic and diastolic blood pressures were measured 3 times using the automatic Blood Pressure monitor and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit. The difference of the msDBP at baseline from the msDBP at 8 weeks was calculated using an Analysis of Covariance (ANCOVA) model with baseline as a covariate and treatment and region as two factors.
Time Frame: Baseline, End of Study (Week 8)
Population: Full Analysis Set (all randomized patients who received study drug). Three patients (1 in Aliskiren 300 mg/Amlodipine 10 mg group and 2 in the Aliskiren 300 mg/Amlodipine 5 mg group were excluded from the analysis due to lack of post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 281 | 274 | 260
mm Hg | -13.07 (0.463) | -10.54 (0.467) | -5.84 (0.480)

2. Secondary Outcome: Change From Baseline to End of Study in the Mean Sitting Systolic Blood Pressure (msSBP)
Description: After the patient had been sitting for 5 minutes, systolic and diastolic blood pressures were measured 3 times using the automatic Blood Pressure monitor and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit. The difference of the msSBP at baseline from the msSBP at 8 weeks was calculated using an ANCOVA model with baseline as a covariate and treatment and region as two factors.
Time Frame: Baseline, End of Study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 281 | 274 | 260
mm Hg | -18.04 (0.780) | -14.43 (0.788) | -6.42 (0.809)

3. Secondary Outcome: Number of Participants With Serious Adverse Events and Adverse Events
Description: The number of participants with any Serious Adverse Event and the number of participants with Adverse Events in any system organ class.
  Additional information about Adverse Events can be found in the Adverse Event Section.
Time Frame: 8 weeks
Population: Safety Population consisted of all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 282 | 276 | 260
participants
  Serious Adverse Events | 3 | 4 | 1
  Adverse Events | 85 | 80 | 59

4. Secondary Outcome: Percentage of Participants Achieving Blood Pressure Control
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using the automatic Blood Pressure monitor and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit.
  Blood Pressure control was defined as having a mean sitting Diastolic Blood Pressure <90 and a mean sitting Systolic Blood Pressure <140.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 281 | 274 | 260
Percentage of participants | 65.5 | 56.5 | 31.5

5. Secondary Outcome: Percentage of Participants Achieving a Diastolic Blood Pressure Response
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using the automatic Blood Pressure monitor and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit.
  A Diastolic Blood Pressure Response was defined as a mean sitting Diastolic Blood Pressure (msDBP) <90 mmHg or a ≥ 10 mmHg reduction in msDBP from baseline.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 281 | 274 | 260
Percentage of participants | 83.6 | 77.7 | 51.5

6. Secondary Outcome: Percentage of Participants Achieving a Systolic Blood Pressure Response
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using the automatic Blood Pressure monitor and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit.
  A Systolic Blood Pressure Response was defined as a mean sitting Systolic Blood Pressure (msSBP) <140 mmHg or a ≥ 20 mmHg reduction in msSBP from baseline.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Number analyzed (Participants) | 281 | 274 | 260
Percentage of participants | 77.2 | 69.7 | 43.8

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Safety set (all patients who received at least 1 dose of double-blind study drug).
Arm/Group | Aliskiren 300 mg/Amlodipine 10 mg | Aliskiren 300 mg/Amlodipine 5 mg | Aliskiren 300 mg
Serious Adverse Events (participants affected / at risk) | 3/282 | 4/276 | 1/260
Other Adverse Events (participants affected / at risk) | 26/282 | 6/276 | 1/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg/Amlodipine 10 mg (N=282) | Aliskiren 300 mg/Amlodipine 5 mg (N=276) | Aliskiren 300 mg (N=260)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg/Amlodipine 10 mg (N=282) | Aliskiren 300 mg/Amlodipine 5 mg (N=276) | Aliskiren 300 mg (N=260)
Oedema peripheral (General disorders) | 26 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.